CLINICAL TRIAL: NCT05653245
Title: The Use of Adhesion Molecule Loaded Hydrogel With Minimally Invasive Surgical Technique in Treatment of Periodontal Intrabony Defect (Randomized Clinical and Biochemical Study)
Brief Title: The Use of Adhesion Molecule Loaded Hydrogel With Minimally Invasive Surgical Technique in Treatment of Periodontal Intrabony Defect
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, shaimaa hamdy, periodontist, Minia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: periodontal regeneration
Record Dates: First submitted 2022-11-29; First posted 2022-12-16 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-11

CONDITIONS: Periodontitis
Keywords: adhesion molecule; intrabony defect; hydrogel; Minimally invasive surgical technique
MeSH Terms: conditions — Periodontitis | interventions — arginyl-glycyl-aspartic acid

STUDY DESIGN:
Intervention Model Description: The total of 45 infra-bony defects were randomly divided into 3 equal groups (n=15 each) by simple randomization and all surgeries were done by the same periodontist (Sh.H):
  * Group 1: Fifteen intra-bony defect sites were treated with modified minimally invasive surgical technique M-MIST alone.
  * Group 2: Fifteen intra-bony defect sites were treated with M-MIST and placebo hydrogel injection.
  * Group3: Fifteen intra-bony defect sites were treated with M-MIST and RGD peptide hydrogel injection.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Placebo Comparator): Fifteen periodontitis patients will receive Phase I therapy, reevaluation after four weeks with modified minimally invasive surgical technique (M-MIST) alone
  Interventions: Drug: RGD Peptide
- Group 2 (Placebo Comparator): Fifteen periodontitis patients will receive Phase I therapy, reevaluation after four weeks with (M-MIST) and hydrogel injection
  Interventions: Drug: RGD Peptide
- Group 3 (Active Comparator): Fifteen periodontitis patients will receive Phase I therapy, reevaluation after four weeks with (M-MIST) and RGD peptide hydrogel.
  Interventions: Drug: RGD Peptide

INTERVENTIONS:
Drug: RGD Peptide — adhesion molecules

SUMMARY:
Primary aim of the study is to evaluate efficacy of RGD adhesion molecule loaded hydrogel with minimally invasive surgical technique in treatment of periodontal intrabony defect at baseline and 6months. Secondary outcome is the biochemical evaluation to detect bone morphogenetic proteins level

DETAILED DESCRIPTION:
Periodontitis is a multifactorial inflammatory disease associated with dysbiotic plaque biofilms and characterized by clinical attachment loss caused by the destruction of the periodontal ligament and loss of supporting bone. One of periodontal therapy goals is regeneration of the lost periodontal attachment apparatus.

. To regenerate healthy periodontal tissue, various clinical techniques were developed to prevent downward epithelial migration and promote periodontal tissue regeneration by the remaining periodontal ligament (PDL) cells or osteoblasts such as open flap debridement (OFD), natural or synthetic filling materials and guided tissue regeneration (GTR).

. Tissue engineering has become one of the most commonly used approaches for bone tissue reconstruction and regeneration, injectable hydrogels have attracted the attention of biomaterials scientists for bone tissue-engineering applications, because they can replace regenerative surgery with a minimally invasive injection method and can form any desired shape, to match irregular defects. Various injectable hydrogels with good moldability and 3D structures have been widely investigated for use in bone tissue engineering.

. Recently a variety of bioactive peptides have been studied and applied for the promotion of bone regeneration to repair local bone defects or treat other bone diseases including extracellular matrix (ECM)- derived peptides, bone morphogenetic proteins (BMPs)-derived peptides and others.

. The arginyl-glycyl-aspartic acid (RGD) peptide is one of bioactive peptides which is the cardinal integrin-binding domain and presents in many extracellular matrix proteins, such as fibronectin and vitronectin. As a part of cell surface signalling, RGD peptide can enhance the expression of osteocalcin (OCN), osteopontin (OPN) and BMP to ensure osteoblast proliferation, differentiation and mineralization.

. The induction of bone depending on the concentration of BMPs which considered important bone biological factors that play essential roles in osteogenesis. BMPs are members of secreted signaling proteins that belong to transforming growth factor beta (TGF-β) superfamily. It has been demonstrated that BMPs induce bone formation by differentiating mesenchymal stem cells to osteoblastic cells

ELIGIBILITY:
Inclusion Criteria:

- Patients with diagnosis of periodontitis (stage III or IV and grade B or C) according to new American Academy of Periodontology classification (Tonetti et al., 2018a) (Nguyen et al., 2021).

* Selected patients of both sexes were 20-55 years old.
* All single and multiple rooted teeth in both maxilla and mandible.
* Presence of interdental periodontal pocket with intrabony defect.
* Patients were free from any systemic diseases that could alter their periodontal status, complicate the surgical treatment, or affect healing according to Modified Cornell Index (Abramson, 1966).
* No antibiotics or any medications that affect bone or soft tissue condition were taken during the last six months.

Exclusion Criteria:

* Patients who received regenerative periodontal therapy last 6 months before the initial examination.

  * Pregnant or lactating females.
  * Smokers were not included as participants in this study.
  * Patients not committed to oral hygiene after the re-evaluation of phase I therapy.
  * Teeth with mobility more than Grade I.
  * Third molars.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-02-05 (Actual); Study Completion 2022-09-09 (Actual)

PRIMARY OUTCOMES:
evaluation of intrabony component dimension component dimension | 6 months follow up
  evaluation of intrabony component dimension (defect base fill) length measured by millimeters
evaluation of intrabony component dimension | 6 months follow up
  crestal bone level length measured by millimeters
evaluation of intrabony component dimension | 6 months follow up
  defect width measured by millimeters

SECONDARY OUTCOMES:
evaluate the clinical parameters attachment gain | 6 months follow up
  The secondary outcomes were to evaluate the clinical attachment gain measured by millimeters
evaluate the clinical parameters | 6 months follow up
  pocket depth reduction measured by millimeters
evaluate the clinical parameters | 6 months follow up
  full-mouth plaque index, full mouth sulcular bleeding index by score

OTHER OUTCOMES:
biochemical evaluation | 1, 7,14 days follow up
  measure bone morphogenetic protein level in gingival crevicular fluid by ELIST test

CONTACTS AND LOCATIONS:
Locations (1):
- Shaimaa Hamdy, Minya, Egypt

IPD SHARING:
Plan to Share IPD: No